CLINICAL TRIAL: NCT00165776
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel, Group Dose-Response, Study of E2014 in Patients WIth Spasmodic Torticollis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2014-J081-131
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-02

CONDITIONS: Cervical Dystonia; Spasmodic Torticollis
MeSH Terms: conditions — Torticollis | interventions — rimabotulinumtoxinB

INTERVENTIONS:
Drug: BOTULINUM TOXIN TYPE B

SUMMARY:
To evaluate efficacy and safety of E2014 (2500U, 5000U, 10000U, placebo) in a multicenter, randomized, double-blind, parallel group comparative study by intramuscularly administering to patients with spasmodic torticollis. Primary endpoint for efficacy evaluation is changes in TWSTRS total scores from baseline measured at Week 4 and the clinical recommended dose will be examined with Williams multiple comparison. For safety evaluation, an inter group comparison (active drug and placebo) will be performed mainly focusing on incidence of adverse events, adverse drug reactions, and abnormal changes in laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can give written informed consent and aged between greater than or equal to 20 years and less than 75 years at the time of obtaining prior consent (irrespective of gender).
* Patients with dystonic symptoms at least 2 or more lesions in the following cervical muscles.
* Sternocleidomastoid
* Scalenus complex (scalenus anterior, scalenus medius, and scalenus posterior)
* Trapezius
* Levator scapulae
* Splenius capitis
* Semispinalis capitis
* Patients who persistently have symptoms in the above (2) for 1 year or longer.
* Patients weighing greater than or equal to 40 kg.
* Patients whose TWSTRS total score at baseline is greater than or equal to 20.
* Patients whose TWSTRS-severity score at baseline is greater than or equal to 10.
* Patients whose TWSTRS-disability score at baseline is greater than or equal to 3.
* Patients whose TWSTRS-pain score at baseline is greater than or equal to 1.
* Patients who are judged to be eligible for study entry by the investigator or subinvestigator based on their physical and neurological findings, laboratory parameters, and ECG results.

Exclusion Criteria:

* Patients who are botulinum toxin-resistant in previous exposures (primary no-responder*)

  *If patients who were once responder to botulinum toxin treatment but thereafter became non-responder can be included in this study.
* Patients whose passive range of motion in the neck is significantly narrowed due to cervical contracture or spondylosis.
* Patients having only pure retrocollis- or anterocollis-associated symptoms.
* Patients who received botulinum toxin agents within 4 months prior to study treatment of E2014, or those who show carry-over effect of previous treatment with botulinum toxin at the time of starting study administration even though the previous treatment was given 4 months or earlier.
* Patients who were treated with narcotics or antibiotics that may potentiate effects of muscle relaxation (spectinomycin hydrochloride preparations, aminoglycosides, polypeptides, tetracyclines, lincomycins) within 4 months prior to study treatment.
* Patients who started or altered the dose levels of the following agents (musculoskeletal relaxants, antispasm drugs, strong tranquilizers, benzodiazepines including similar drugs, anticholinergic drugs, antiparkinsonian drugs, antidepressants) within 4 weeks prior to study treatment.
* Patients who received medical care(s) other than pharmacotherapies (surgical interventions, MAB, acupuncture, relaxation, etc.) prior to study treatment showing carry-over effect of these cares or unstable condition at the time of starting study treatment.
* Patients who have a history of myectomy or neurectomy in the neck and/or shoulder.
* Patients who have a history of hypersensitivity to E2014's ingredients (botulinum toxin type B, human serum albumin, sodium succinate buffer solution), or other type of botulinum toxins.
* Patients with complication(s) or history of serious neurological or musculoskeletal disease (myasthenia, amyotrophic lateral sclerosis, etc.), cardiovascular disease (acute myocardial infarction, etc.), respiratory disease (COPD, etc.), renal disease (acute or chronic renal failure, etc.), hepatic disease (cirrhosis, etc.), gastrointestinal disease (paralytic ileus, etc.), dermatological disease (toxic epidermal necrosis, etc.), psychiatric disease (schizophrenia, alcohol or drug dependence, etc.), hematological disease (aplastic anemia, etc.), and/or infectious disease (hepatitis, syphilis, AIDS, etc.).
* Patients with complication or history of malignant tumor(s).
* Patients who participated in another clinical study within 30 days prior to obtaining informed consent for this study.
* Women of pregnant, childbearing potential, childbearing intension during the study period, or lactating.
* Others who are judged to be ineligible for study entry by the investigator or subinvestigator

Ages: 20 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2004-06; Primary Completion 2006-05 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Japan (19):
  - Ichihara, Chiba
  - Kitakyushu, Fukuoka
  - Sapporo, Hokkaido
  - Kagoshima, Kagoshima-ken
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Kyoto, Kyoto
  - Matsumoto, Nagano
  - Kashihara, Nara
  - Moriguchi, Osaka
  - Osaka, Osaka
  - Sakai, Osaka
  - Saitama, Saitama
  - Tokorozawa, Saitama
  - Hamamatsu, Shizuoka
  - Tokushima, Tokushima
  - Bunkyo-ku, Tokyo
  - Meguro-ku, Tokyo
  - Shinjuku-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 130 patients (33 of the placebo group, 34 of the 2500U group, 32 of the 5000U group, and 31 of the 10000U group) received study treatment, but after randomization, 3 patients (2 of the placebo group and 1 of the 5000U group) had no treatment. The reason was that 2 of them requested withdrawal from the study and 1 ceased to return for visits.
Groups:
- Placebo: placebo/ 2 mL was intramuscularly injected to cervical muscles as a single dose
- E2014 2,500 U: 2,500 U/2 mL was intramuscularly injected to cervical muscles as a single dose
- E2014 5,000 U: 5,000 U/2 mL was intramuscularly injected to cervical muscles as a single dose
- E2014 10,000 U: 10,000 U/2 mL was intramuscularly injected to cervical muscles as a single dose
Period: Overall Study
Arm/Group | Placebo | E2014 2,500 U | E2014 5,000 U | E2014 10,000 U
Started | 35 | 34 | 33 | 31
Completed | 31 | 33 | 31 | 29
Not Completed | 4 | 1 | 2 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 2 | 0
Not completed — Worsening of Cervical Dystonia | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: After randomized to the treatment groups, 3 patients (2 of the placebo group and 1 of the 5000U group) had no treatment. The reason was that 2 of them requested withdrawal from the study and 1 ceased to return for visits.
Groups:
- Placebo: placebo/ 2 mL was intramuscularly injected to cervical muscles as a single dose. Two subjects from the placebo group did not receive treatment after randomization.
- E2014 5,000 U: 5,000 U/2 mL was intramuscularly injected to cervical muscles as a single dose. One subject from the 5,000 U/2 mL did not receive treatment after randomization.
- Total: Total of all reporting groups
Arm/Group | Placebo | E2014 2,500 U | E2014 5,000 U | E2014 10,000 U | Total
Number analyzed (Participants) | 33 | 34 | 32 | 31 | 130
Age, Customized [Number; unit: Participants]
  Less than 40 years | 10 | 11 | 10 | 8 | 39
  40 to less than 60 years | 12 | 8 | 18 | 13 | 51
  Greater than or equal to 60 years | 11 | 15 | 4 | 10 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 15 | 14 | 52
  Male | 21 | 23 | 17 | 17 | 78
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 33 | 34 | 32 | 31 | 130

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change From Baseline in Patient Global Assessment - Visual Analog Scale (PtGA-VAS) at Week 4 After Treatment
Description: Change from Baseline in PtGA-VAS is computed as Week 4 value minus baseline value. A negative value in change from baseline indicates an improvement. Participants answered: "Considering all the ways your cervical dystonia affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm VAS, where 0 mm = very well and 100 mm = very poorly.
Time Frame: Baseline, Week 4
Population: FAS
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Placebo | E2014 2,500 U | E2014 5,000 U | E2014 10,000 U
Number analyzed (Participants) | 33 | 34 | 32 | 31
Millimeters | -0.4 (3.2) | 11.9 (2.6) | 9.9 (3) | 13.3 (3)

2. Secondary Outcome: Mean Change From Baseline in Physician Global Assessment Disease Assessment - Visual Analog Scale (PGA-VAS) at Week 4 After Treatment
Description: Change from Baseline in PGA-VAS (0 to 100 mm visual analog scale, 0 being no symptoms and 100 being severe symptoms) is computed as Week 4 value minus baseline value. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline, Week 4
Population: FAS
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Placebo | E2014 2,500 U | E2014 5,000 U | E2014 10,000 U
Number analyzed (Participants) | 33 | 34 | 32 | 31
Millimeters | 2 (2.2) | 10.6 (2.9) | 11.2 (2.6) | 16.9 (2.8)

3. Primary Outcome: Mean Change From Baseline in the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) -Total Score at Week 4 After Treatment
Description: The TWSTRS-Total score is the sum of scores of the three components of the scale:
  * TWSTRS-Severity score which ranges from 0 (=absence of severity) to 35 points (=maximum severity)
  * TWSTRS-Pain score which ranges from 0 (=no pain) to 20 (=maximum pain)
  * TWSTRS-Disability score which ranges from 0 (=no disability) to 30 (=maximum disability).
  The TWSTRS total score ranges from 0 (=best value) to 85 (=worst value). The change from baseline was calculated as the score at the corresponding visit minus the baseline score.
Time Frame: Baseline, Week 4
Population: Full Analysis Set (FAS) population: All subjects who received study treatment
Measure: Mean (Standard Error); unit: Points on a Scale
Arm/Group | Placebo | E2014 2,500 U | E2014 5,000 U | E2014 10,000 U
Number analyzed (Participants) | 33 | 34 | 32 | 31
Points on a Scale | 3 (1.3) | 8.9 (1.8) | 7.6 (1.6) | 10.5 (1.6)

4. Secondary Outcome: Mean Change From Baseline in the TWSTRS - Functional Disability Score at Week 4 After Treatment
Description: TWSTRS-Disability score which ranges from 0 (=no disability)to 30 (=maximum disability). The change from baseline was calculated as the score at the corresponding visit minus the baseline score.
Time Frame: Baseline, Week 4
Population: FAS
Measure: Mean (Standard Error); unit: Points on a Scale
Arm/Group | Placebo | E2014 2,500 U | E2014 5,000 U | E2014 10,000 U
Number analyzed (Participants) | 33 | 34 | 32 | 31
Points on a Scale | 0.6 (0.7) | 2.5 (0.6) | 1.9 (0.8) | 3.1 (0.5)

5. Secondary Outcome: Mean Change From Baseline in the TWSTRS - Pain Score at Week 4 After Treatment
Description: TWSTRS-Pain score which ranges from 0 (=no pain) to 20 (=maximum pain). The change from baseline was calculated as the score at the corresponding visit minus the baseline score.
Time Frame: Baseline, Week 4
Population: FAS
Measure: Mean (Standard Error); unit: Points on a Scale
Arm/Group | Placebo | E2014 2,500 U | E2014 5,000 U | E2014 10,000 U
Number analyzed (Participants) | 33 | 34 | 32 | 31
Points on a Scale | 0.8 (0.4) | 2.9 (0.7) | 2 (0.7) | 2.7 (0.7)

6. Secondary Outcome: Mean Change From Baseline in the TWSTRS - Severity Score at Week 4 After Treatment
Description: TWSTRS-Severity score which ranges from 0 (=absence of severity) to 35 points (=maximum severity). The change from baseline was calculated as the score at the corresponding visit minus the baseline score.
Time Frame: Baseline, Week 4
Population: FAS
Measure: Mean (Standard Error); unit: Points on a Scale
Arm/Group | Placebo | E2014 2,500 U | E2014 5,000 U | E2014 10,000 U
Number analyzed (Participants) | 33 | 34 | 32 | 31
Points on a Scale | 1.6 (0.6) | 3.5 (0.8) | 3.7 (0.7) | 4.7 (0.8)

7. Secondary Outcome: Mean Change From Baseline in Patient Pain Assessment (VAS) at Week 4 After Treatment
Description: Change from Baseline in Patient's Pain Assessment-VAS is computed as Week 4 value minus baseline value. A negative value in change from baseline indicates an improvement. The patient's assessment of pain was performed using a 100 mm VAS)ranging from no pain (0) to unbearable pain (100). The distance in mm from the left edge of the scale was measured. A negative change from Baseline score indicates improvement in pain intensity.
Time Frame: Baseline, Week 4
Population: FAS
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Placebo | E2014 2,500 U | E2014 5,000 U | E2014 10,000 U
Number analyzed (Participants) | 33 | 34 | 32 | 31
Millimeters | -6.6 (4.1) | -15 (4.5) | -13.4 (4.7) | -8.7 (4.4)

ADVERSE EVENTS:
Time Frame: Baseline to last observation carried forward
Description: 130 patients (33 of the placebo group, 34 of the 2500U group, 32 of the 5000U group, and 31 of the 10000U group) received study treatment, but after randomization, 3 patients (2 of the placebo group and 1 of the 5000U group) had no treatment. The reason was that 2 of them requested withdrawal from the study and 1 ceased to return for visits.
Arm/Group | Placebo | E2014 2,500 U | E2014 5,000 U | E2014 10,000 U
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34 | 0/32 | 2/31
Other Adverse Events (participants affected / at risk) | 9/33 | 3/34 | 4/32 | 7/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=33) | E2014 2,500 U (N=34) | E2014 5,000 U (N=32) | E2014 10,000 U (N=31)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | E2014 2,500 U (N=34) | E2014 5,000 U (N=32) | E2014 10,000 U (N=31)
Nasopharyngitis (Infections and infestations) | 9 | 2 | 4 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 3 | 7
Thirst (General disorders) | 1 | 1 | 1 | 6
Headache (Nervous system disorders) | 1 | 1 | 1 | 3
Injection Site Pain (General disorders) | 2 | 0 | 2 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 2 | 0 | 2
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Glucose Urine Present (Investigations) | 0 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No